CLINICAL TRIAL: NCT07000721
Title: Research on New Intelligent Diagnosis and Treatment Technologies for Early Lung Cancer Based on Multimodal Imaging Bronchoscopy Navigation
Brief Title: Research on New Diagnosis and Treatment Technologies for Early Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jisong Zhang (Other)
Responsible Party: Sponsor-Investigator, Jisong Zhang, Doctor of Medicine, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SirRRSH2024-1000
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer, Peripheral Pulmonary Nodules
Keywords: Lung cancer; peripheral pulmonary nodules; AI-constructed airway tree navigation system; diagnosis; effectiveness and safety
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New navigation system group (Experimental): The new AI-constructed airway tree navigation system (SARS-pro) was used for preoperative navigation path planning. The SARS-pro navigation system was independently developed by the research group based on a conventional augmented reality optical navigation system (LungPro; Bronchus Company).
  Interventions: Diagnostic Test: Preoperative navigation path planning using the SARS-pro navigation system
- Old navigation system group (Active Comparator): Preoperative navigation path planning was performed using the old VBN system (LungPro; Bronchus Company).
  Interventions: Diagnostic Test: Preoperative navigation path planning using the VBN navigation system

INTERVENTIONS:
Diagnostic Test: Preoperative navigation path planning using the SARS-pro navigation system — The SARS-pro navigation system was used for preoperative navigation path planning for tracheoscopic biopsies in the new navigation system group (patients with suspected lung cancer).
  Arms: New navigation system group
Diagnostic Test: Preoperative navigation path planning using the VBN navigation system — The VBN navigation system was used for preoperative navigation path planning for tracheoscopic biopsies in the old navigation system group (patients with suspected lung cancer).
  Arms: Old navigation system group

SUMMARY:
To verify the clinical effectiveness and safety of the airway tree navigation system constructed by artificial intelligence (AI) in the navigation diagnosis of peripheral pulmonary nodules (PPLs).

DETAILED DESCRIPTION:
Early diagnosis and treatment of lung cancer is of great significance, in which navigated tracheoscopic biopsy is an important tool for confirming the diagnosis of early lung cancer. Conventional navigation software realizes airway reconstruction and guides biopsy by recognizing differences in HU values on computed tomography scans. It is difficult for conventional navigation software to recognize the reconstruction due to the special characteristics of small airways that are susceptible to interference and collapse. Therefore, an AI deep learning approach can realize accurate construction of small airways and guide accurate biopsy. This study intends to validate the clinical effectiveness and safety of the AI-constructed airway tree navigation system in the navigational diagnosis of peripheral pulmonary nodules (PPLs).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above.
2. Patients with one or more peripheral lung nodules suspected to be lung cancer or poorly absorbing lesions on conventional anti-infective therapy.
3. Patients with nodule diameters ≤30 mm (diameters mentioned in the text are the average of the maximum and minimum diameters).
4. The nodules were pure ground glass nodules, partially solid nodules, or solid nodules.
5. The nodule is surrounded by lung parenchyma and is not visible in the bronchial lumen above the segment.

Exclusion Criteria:

1. Preoperative judgment that it is difficult for the patient to benefit from bronchoscopic biopsy (e.g., high risk of bleeding due to perivascular encasement of the lesion, difficulty in reaching the airway adjacent to the lesion due to previous lung surgery, etc.).
2. Those with incomplete clinical data.
3. Those with missing visits after biopsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic positive yield | One month after the patients were enrolled
  After biopsy by navigational bronchoscopy, the biopsy tissue was tested for lung cancer pathology. A positive diagnosis was defined when the pathology report was a neoplastic lesion (benign or malignant tumor). A positive diagnosis was also made if the pathology report was a granulomatous lesion (with tuberculosis or fungus). If the pathology was reported as an inflammatory cell infiltration or other non-specific inflammation in the lungs, the subject underwent another pathology biopsy after at least 3 months of follow-up to rule out false-positive results due to a change in the site of the lesion.

SECONDARY OUTCOMES:
Adverse events | 3 days after navigational tracheoscopic biopsy
  Patients underwent a follow-up period of 3 days after navigational tracheoscopic biopsy, and subjects were followed for adverse events such as hemoptysis, pneumothorax, and mediastinal emphysema.

CONTACTS AND LOCATIONS:
Overall Officials: Enguo Chen, MD, Study Director — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT07000721/Prot_SAP_ICF_000.pdf